CLINICAL TRIAL: NCT01186510
Title: Lung Perfusion With Oxygenated Blood During Aortic Clamping
Acronym: PulPer-001-Sch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, Head Cardiovascular Research, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PulPer-001-Sch
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Postoperative Pulmonary Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung perfusion (Experimental)
  Interventions: Procedure: lung perfusion
- no lung perfusion (Active Comparator)
  Interventions: Procedure: no lung perfusion

INTERVENTIONS:
Procedure: lung perfusion — see literature of proceeding
  Arms: Lung perfusion
Procedure: no lung perfusion — see literature of proceeding
  Arms: no lung perfusion

SUMMARY:
Pulmonary dysfunction presumably linked to an inflammatory response is frequent after cardiac operations using cardiopulmonary bypass (CPB) and pulmonary hypoperfusion.

Aim of the study: To evaluate the protective effect of continuous pulmonary perfusion with oxygenated blood during aortic crossclamping on the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 ys
* Cardiopulmonary bypass procedure
* FEV1 <80%
* COPD >II

Exclusion Criteria:

* Emergency cases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Inflammatory marker | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Goethe University, Frankfurt am Main, Germany

REFERENCES:
- [Derived] Kiessling AH, Guo FW, Gokdemir Y, Thudt M, Reyher C, Scherer M, Beiras-Fernandez A, Moritz A. The influence of selective pulmonary perfusion on the inflammatory response and clinical outcome of patients with chronic obstructive pulmonary disease undergoing cardiopulmonary bypass. Interact Cardiovasc Thorac Surg. 2014 Jun;18(6):732-9. doi: 10.1093/icvts/ivu062. Epub 2014 Mar 14. PMID 24632426